CLINICAL TRIAL: NCT01949389
Title: Piloting an Internet-based Therapy for Insomnia in a Population of Veterans With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Rosenheck, Senior Health Serivces Investigator, VA Connecticut Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01633
Record Dates: First submitted 2013-09-05; First posted 2013-09-24 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-based Cognitive Behavioral Therapy for Insomnia (Experimental): This is an internet-based Cognitive Behavioral treatment for insomnia. It is accessed via a computer with an internet connection and consists of 7 modules, homework, and a daily sleep log. The intervention is self administered.
  Interventions: Behavioral: Internet-based Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioral Therapy for Insomnia — This is an internet-based Cognitive Behavioral treatment for insomnia. It is accessed via a computer with an internet connection and consists of 7 modules, homework, and a daily sleep log. The intervention is self administered.

SUMMARY:
The purposes of this study is to examine the feasibility of implementing an internet-based treatment for insomnia among veterans with substance use disorders, some with co-morbid serious mental illness, and to develop potential methods to support and encourage veterans while they self-administer this treatment. Our hypotheses are that the implementation of an internet-based therapy will be feasible and that a method of support can be devised, and tested in the future.

ELIGIBILITY:
Inclusion Criteria:

* Inability to sleep within 30 minutes of going to bed or awakening during the night for 30 minutes for greater than or equal to 3 days per week
* Above Criteria occurring every week for greater than or equal to 3 months
* At least one symptom of daytime impairment: (reduced motivation, sleepiness, fatigue, lack of concentration, performance at home, work, social life, relationships impaired)
* Able to provide valid consent
* Willing to participate in an internet-based cognitive behavioral therapy for insomnia
* English speaking

Exclusion Criteria:

* Self-reported or provider diagnosed sleep apnea or related nighttime respiratory problem, restless legs syndrome or related nighttime movement disorder
* Acute psychiatric decompensation requiring inpatient admission or emergency department services within the last month (suicidality, homicidally, mania, psychotic decompensation)
* Current treatment or treatment within the last month for opiate addiction with methadone maintenance or buprenorphine.
* Has a conservator E. Shift work interfering with the establishment of regular sleep patterns F. Previous or ongoing cognitive behavioral therapy for insomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 Individuals were recruited between October 2013 and May 2014.
Pre-assignment Details: A single subject completed informed consent procedures and signed the informed consent document, but then was found not to meet exclusion criteria on review of the medical record. The individual was disenrolled.
Period: Overall Study
Arm/Group | Internet-based Cognitive Behavioral Therapy for Insomnia
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Veterans recieving care at the VA Connecticut out patient Substance Use Disorders Clinic
Arm/Group | Internet-based Cognitive Behavioral Therapy for Insomnia
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — gender
  Participants
    Female | 6
    Male | 45
Race/Ethnicity, Customized [Number; unit: participants]
  White | 27
  African American | 19
  Other Race/Ethnicity | 5
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (Total), Change From Baseline to Follow-up
Description: Insomnia Severity Index (Total) following completion of the intervention (expected average of 7 weeks)
  The Insomnia Severity Index is a self-report seven-item measure that targets the subjective symptoms and functional consequences of insomnia as well as the degree of concerns or distress caused by those difficulties, and corresponds to the diagnostic criteria of insomnia. Scores range from 0-28, higher scores indicate more severe insomnia, and scores ≥15 suggest moderate to severe insomnia.
Time Frame: pre-intervention, intervention completion (expected average of 7 weeks)
Population: The number of individuals provided access to the program and reporting baseline and follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Cognitive Behavioral Therapy for Insomnia
Number analyzed (Participants) | 45
units on a scale | 6.3 (2.3)

2. Primary Outcome: Completion of All 7 Modules of the Intervention
Description: Participants will be followed for the duration of the intervention (7 individual modules, completed weekly, for an expected average of 7 weeks). Outcome measure will be characterized as the number completing all 7 modules of the program (dichotomous variable).
  The intervention is a 7-week, self-administered course accessed via the Internet that includes instruction on psycho-education, stimulus control, relaxation training, sleep restriction, medication tapering, cognitive distortions, and mindfulness integrated into each module. Homework is assigned after each module. Participants are instructed to complete the sleep diary included in the program daily while participating in the program.
Time Frame: on average 7 weeks
Measure: Number; unit: participants
Arm/Group | Internet-based Cognitive Behavioral Therapy for Insomnia
Number analyzed (Participants) | 51
participants | 21

ADVERSE EVENTS:
Arm/Group | Internet-based Cognitive Behavioral Therapy for Insomnia
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes